CLINICAL TRIAL: NCT00277290
Title: A Phase 2 Study of XL999 Administered Intravenously to Subjects With Recurrent Ovarian Cancer
Brief Title: Study of XL999 in Patients With Previously Treated Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to cardiac toxicities in the subjects
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-202
Expanded Access: Available
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Ovarian Cancer
Keywords: Cancer; Recurrent; Platinum-resistant; Platinum-sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — Treatment was administered on an outpatient basis. XL999 was administered at 2.4 mg/kg as a 4 hour intravenous (IV) infusion. Subjects received a XL999 infusion once a week for 8 weeks of treatment unless drug-related toxicity required a dosing delay

SUMMARY:
This clinical trial is being conducted at multiple sites to evaluate the activity, safety, and tolerability of XL999 when given weekly to patients with ovarian cancer that has previously been treated with platinum-based chemotherapy. XL999 is a small molecule inhibitor of multiple kinases including VEGFR, PDGFR, FGFR, FLT-3, and Src, which are involved in tumor cell growth, formation of new blood vessels (angiogenesis), and metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with a histologically confirmed diagnosis of metastatic ovarian cancer
* Measurable disease according to Response Criteria for Solid Tumors (RECIST)
* Prior treatment with platinum-based therapy
* Platinum-sensitive or platinum-resistant disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of ≥3 months
* Adequate organ and marrow function
* Signed informed consent
* No other malignancies within 5 years

Exclusion Criteria:

* Radiation to ≥25% of bone marrow within 30 days of XL999 treatment
* Use of an investigational drug or cytotoxic chemotherapy within 30 days of XL999 treatment
* Prior anticancer therapy targeting VEGF (eg, bevacizumab, sorafenib, or sunitinib)
* More than two prior systemic non-platinum cytotoxic chemotherapy regimens
* Subject has not recovered to grade ≤1 or to within 10% of baseline from adverse events due to other medications administered >30 days prior to study enrollment
* History of or known brain metastases, current spinal cord compression, or carcinomatous meningitis
* Uncontrolled and/or intercurrent illness
* Patients who are pregnant or breastfeeding
* Known human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Response rate | Inclusion until disease progression
Safety and tolerability | Inclusion until 30 days post last treatment

SECONDARY OUTCOMES:
Progression-free survival | Inclusion until disease progression
Duration of response | Inclusion until disease progression
Overall survival | inclusion until 180-Day Follow-up after last treatment or death
Pharmacokinetic (PK) and pharmacodynamics (PD) parameters | Samples will be collected pre-dose and immediatelyat the end of infusion for the 8-week Study Treatment Period for subjects in the second stage of the study

CONTACTS AND LOCATIONS:
Overall Officials: Lynne A. Bui, MD, Study Director — Exelixis
Locations (9):
- United States (9):
  - California Cancer Care, Inc., Greenbrae, California
  - Hematology/Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Ltd, Joliet, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bradley Cohen, New City, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York